CLINICAL TRIAL: NCT03665623
Title: A Prospective Multi-center Study on the Prediction of Preeclampsia by Comprehensive Markers in Early Pregnancy.
Brief Title: Prediction of Preeclampsia by Comprehensive Markers.
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: preeclampsia prediction study
Record Dates: First submitted 2018-06-12; First posted 2018-09-11 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Pre-Eclampsia
Keywords: preeclampsia prediction; competing risk model; 11~13+6 gestational weeks
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — maternal serum samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preeclampsia is one of the most serious complications in pregnancy that causes maternal death and preterm delivery. Series studies has show that the competing risk model developed by the Fetal Maternal FouNdation in early pregnancy has the potential to predict preeclampsia effectively but has show crowd difference. We aim to evaluate the performance of various screening model based on FMF model in Chinese population.

DETAILED DESCRIPTION:
The prospective multi-center observational study aimed to recruit at least 10,000 pregnant woman during the first trimester conducted among 12 medical centers in China. The medical history of each candidate was recorded , blood pressure was measured , blood sample was taken between 11 gestational weeks and 13+6 gestational weeks, to get the PlGF and PAPPA tested. Routine ultrasound was taken with measurement of the uterine artery pulsatility index. The results of the recruited patients were not released to the patients or the doctor. Pregnancy outcome was recorded as to whether the women develop preeclampsia , the SGA babies, or low birth Apgar score and other preeclampsia related adverse maternal and neonatal outcomes. The basic medical information, the mean artery pressure, the PlGF and PAPPA MOM, the UtA PI were used in combination to do the risk stratification, and to develop prediction model for Chinese people.

ELIGIBILITY:
Inclusion Criteria:

1. gestational weeks between 11~13+6
2. agreed to participate the study
3. live fetus at recruitment.

Exclusion Criteria:

1. first obstetric visit beyond 14 gestational weeks
2. artificial abortion or spontaneous abortion before 20 weeks or lost to follow-up.
3. refused to participate the study.
4. fetus with major chromosome or structural abnormality

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — we recruit pregnant women who visit the hospital between gestational weeks 11-13+6 days ,have routine visits and planned delivery in registered hospital,singed agreement to participate the study.
Study Population: we aimed to recruit as many as possible the women without discrimination during the study periods.
Sampling Method: Non-Probability Sample
Enrollment: 11741 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
detection rate of preterm preeclampsia at fixed false positive rate 5%,10%,15%,20% | at delivery and reviewed 60 days postpartum
  PE defined according to the International Society for the Study of Hypertension in Pregnancy and the American College of Obstetricians and Gynecologists.

SECONDARY OUTCOMES:
detection rate of small for gestational neonates at fixed risk cut of defined in primary outcome | at delivery
  defined as birthweight above or below the 90th and 10th centiles of our local population standard chart after adjusting for gender and gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China